CLINICAL TRIAL: NCT04190030
Title: Virginia Commonwealth University Stress Reduction Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Mind & Life Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HM20015897
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Stress
Keywords: Mindfulness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental)
  Interventions: Behavioral: mindfulness training
- Cognitive reappraisal (Active Comparator)
  Interventions: Behavioral: cognitive reappraisal training

INTERVENTIONS:
Behavioral: mindfulness training — Participants will listen to 20-minute lessons each day for 14 days plus complete brief (3 to 10 minute) exercises daily via their personal smartphone. Each course will involve mental exercises to reduce stress in daily life, along with direct instruction from the course leader to help in learning and applying the stress reduction techniques.
  Arms: Mindfulness
Behavioral: cognitive reappraisal training — Participants will listen to 20-minute lessons each day for 14 days plus complete brief (3 to 10 minute) exercises daily via their personal smartphone. Each course will involve mental exercises to reduce stress in daily life, along with direct instruction from the course leader to help in learning and applying the stress reduction techniques.
  Arms: Cognitive reappraisal

SUMMARY:
This research study seeks to understand how stress reduction training influences neural responses (brain activation) and behavior related to stress, including emotions and reactions to social conflict.

DETAILED DESCRIPTION:
The full research project will be conducted over approximately 2-3 weeks, and will consist of two data collection sessions, one before and one after a 14-day stress reduction training course conducted via a smartphone that participants provide. This course entails instructor-facilitated stress reduction exercises previously shown to reduce stress and improve well-being. Participants will be randomly assigned to a mindfulness course or a cognitive reappraisal course. Both of these courses -mindfulness training (MT) and cognitive reappraisal training (RT) - involve expert-facilitated mental wellness techniques. MT emphasizes mindfulness-based techniques to reduce stress and promote wellbeing, whereas CT emphasizes reframing and reappraisal techniques to reduce stress and promote well-being.

ELIGIBILITY:
Inclusion Criteria:

* Stable medication regiment for 8 weeks prior to enrollment if taking antidepressant or anxiolytic medications. (will not be advertised but screened)
* Free of major, uncorrected sensory impairments and cognitive deficits
* Free of a certain psychiatric disorders or history thereof; specifically, a new diagnosis of a (non-acute) medical or psychiatric condition within the last 3 months, report a hospitalization over the last 3 months, report current drug abuse (e.g., recreational drug use, alcohol intake in excess of 2 drinks per day).
* Adults aged 18 - 55 years of age
* Right hand dominant (will not be advertised but screened)
* Personal SmartPhone (Android or iOS operating systems).
* Naive to meditation practice (will not be advertised but screened)
* At least a moderate level of perceived stress (scale score > 5 on the 4-item Perceived Stress Scale (PSS; reflects above-average perceived stress)

Exclusion Criteria:

* left-handed
* are unwilling or unable to complete study assessments or treatments
* report a new diagnosis of a (non-acute) medical or psychiatric condition within the last 3 months
* report a hospitalization over the last 3 months
* report current drug abuse (e.g., recreational drug use, smoke more than � pack per day, alcohol intake in excess of 2 drinks per day)
* are prisoners
* no personal SmartPhone (Android or iOS operating systems)

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Functional near-infrared spectroscopy (fNIRS) hemodynamic signal change | Baseline and 16 weeks
  Proportion of participants who show a statistically significant change in regional specificity, as measured by fNIRS-recorded blood oxygenation representing markers of emotion reactivity and regulation during observation of video stimuli.

SECONDARY OUTCOMES:
Change in anger response | Baseline and 16 weeks
  The Anger subscale of the Discrete Emotions Questionnaire (DEQ) will be used to assess s the extent to which participants experience specific emotions on a scale from 1 (not at all) to 7 (an extreme amount) in response to video stimuli. Lower scores indicate less anger and more emotion downregulation. Higher scores would indicate more anger and less emotion downregulation.
Change in disgust response | Baseline and 16 weeks
  The Disgust subscale of the Discrete Emotions Questionnaire (DEQ) will be used to assess the extent to which participants experience specific emotions on a scale from 1 (not at all) to 7 (an extreme amount) in response to video stimuli. Lower scores indicate less disgust and more emotion downregulation. Higher scores would indicate more disgust and less emotion downregulation.
Change in fear response | Baseline and 16 weeks
  The Fear subscale of the Discrete Emotions Questionnaire (DEQ) will be used to assess the extent to which participants experience specific emotions on a scale from 1 (not at all) to 7 (an extreme amount) in response to video stimuli. Lower scores indicate less fear and more emotion downregulation. Higher scores would indicate more fear and less emotion downregulation.
Change in anxiety response | Baseline and 16 weeks
  The Anxiety subscale of the Discrete Emotions Questionnaire (DEQ) will be used to assess the extent to which participants experience specific emotions on a scale from 1 (not at all) to 7 (an extreme amount) in response to video stimuli. Lower scores indicate less anxiety and more emotion downregulation. Higher scores would indicate more anxiety and less emotion downregulation.
Change in sadness response | Baseline and 16 weeks
  The Sadness subscale of the Discrete Emotions Questionnaire (DEQ) will be used to assess the extent to which participants experience specific emotions on a scale from 1 (not at all) to 7 (an extreme amount) in response to video stimuli. Lower scores indicate less sadness and more emotion downregulation. Higher scores would indicate more sadness and less emotion downregulation.
Change in intergroup attitudes | Baseline and 16 weeks
  The Beliefs about Groups survey will be used to assess explicit intergroup attitudes. Participants answer 4 questions using a scale from 1 to 6. Higher scores indicate poorer attitude outcomes.
Behavioral willingness to participate in a dyad-based future experiment | 16 weeks
  Number of participants who express willingness to participate in a dyad-based future experiment using a scale from 1 to 5. Higher scores indicate greater willingness or preference to participate.

CONTACTS AND LOCATIONS:
Overall Officials: Hadley Rahrig, M.S., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No